CLINICAL TRIAL: NCT07206238
Title: Orbital Vascular Inflammation in Ischemic Optic Neuropathy and Giant Cell Arteritis
Acronym: VISION-GCA
Status: Not yet recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Steffen Hamann, Clinical Professor, Rigshospitalet, Denmark
Other Study IDs: H-25043110
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Giant Cell Arteritis (GCA); Ischemic Optic Neuropathy; NAION - Non-Arteritic Ischemic Optic Neuropathy
Keywords: FDG PET/MRI BB; OCT; Retinal biomarkers; Giant cell arteritis; ischemic optic neuropathy
MeSH Terms: conditions — Giant Cell Arteritis; Optic Neuropathy, Ischemic | interventions — Positron-Emission Tomography; Magnetic Resonance Imaging; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anterior ischemic optic neuropathy (AION): Adults aged 50 years or more with new onset AION, here defined as ipsilateral papilledema, visual impairment (affecting BCVA and/or visual field) and relative afferent pupillary defect (RAPD).
  Interventions: Diagnostic Test: Positron Emission Tomography / Magnetic Resonance Imaging
- Giant cell arteritis (GCA) without GCA-related vision loss: Adults aged 50 years or more, newly diagnosed with GCA (clinically and ultrasound-confirmed), and without permanent or transient loss of vision or double vision.
  Interventions: Diagnostic Test: Positron Emission Tomography / Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Positron Emission Tomography / Magnetic Resonance Imaging — FDG PET/MRI with Black Blood sequences of the head and neck area.
  Other Names: Optical Coherence Tomography; Temporal Artery Ultrasound

SUMMARY:
Giant cell arteritis (GCA) is an inflammation of the blood vessels. A dangerous complication is sudden vision loss due to insufficient blood supply to the optic nerve. However, it is often difficult to distinguish acute vision loss due to GCA from a similar condition of insufficient blood supply to the optic nerve, called NAION. Quick treatment with anti-inflammatory medication is needed in case of GCA to prevent vision loss on the eye and other serious complications. Patients with NAION have no benefit of the medication, but can have serious side effects, why it is very important to differentiate between these conditions.

In this project, the investigators will use FDG PET/MRI with Black Blood (BB) sequences and OCT-imaging to study patients with GCA and/or ischemic optic nerve disease. The investigators will look for signs of inflammation in and around the small vessels of the orbit using PET/MRI and study subtle retinal changes using OCT images.

The investigators want to answer the following research questions:

Do patients with ischemic optic nerve disease and GCA show signs of inflammation in the orbital vessel wall on PET/MRI-scans, that are not present in patients with NAION?

Do GCA patients without vision loss, but with signs of orbital vessel wall inflammation on PET/MRI-scans, have a higher risk of later vision loss than GCA patients without?

Can subtle changes in the retina, detectable through OCT, help distinguish between GCA-related vision loss and NAION?

This will, to our knowledge, be the first study to systematically use FDG PET/MRI BB-scans to illuminate vascular changes in the orbit of patients with GCA and/or ischemic optic nerve disease. The results may improve diagnosis and treatment of GCA and NAION in the future. The investigators hope that this will help prevent blindness and other serious complications in patients with GCA, while also avoiding unnecessary treatments for patients with NAION.

DETAILED DESCRIPTION:
Rationale and problem statement:

Giant cell arteritis (GCA) is an immune-driven inflammatory condition affecting the walls of blood vessels. Untreated, GCA can cause vessel wall thickening severe enough to reduce blood flow to various organs. One of the most feared complications is arteritic anterior ischemic optic neuropathy (A-AION), where the anterior part of the optic nerve loses its blood supply, resulting in sudden and often permanent vision loss.

It is crucial to distinguish A-AION from the much more common non-arteritic AION (NAION), since the correct diagnosis directly determines treatment. High-dose corticosteroids must be started immediately when GCA is suspected, in order to reduce the risk of vision loss in the other eye and other severe complications such as stroke or aortic dissection. In contrast, corticosteroid treatment does not benefit patients with NAION and should be avoided because of its significant short- and long-term side effects. However, it remains clinically very difficult to distinguish between A-AION and NAION, even with current diagnostic tools. Furthermore, fundamental knowledge about the vascular changes underlying ischemic optic neuropathy is still lacking.

Imaging background:

18F-Fluorodeoxyglucose (FDG) is a radiolabeled sugar analogue that highlights areas with increased metabolic activity, including inflammatory processes. Previous studies have shown increased FDG uptake in the walls of large and medium-sized arteries in the trunk and skull of GCA patients, but not in the small orbital vessels that supply the eye and optic nerve. Vessel wall inflammation also causes endothelial leakage and thickening, which can be visualized by Magnetic Resonance Imaging (MRI). Prior studies using orbital MRI with Black Blood (BB) sequences have demonstrated thickening and contrast enhancement of orbital vessels in GCA patients.

In addition, smaller studies suggest that patients with ischemic optic neuropathy may have subtle structural changes in the retina, visible on Optical Coherence Tomography (OCT) scans, with different patterns seen in A-AION versus NAION. The frequency and clinical significance of these changes remain poorly understood.

Study objectives:

The main goal of this project is to investigate orbital vessel inflammation in patients with ischemic optic neuropathy and GCA, specifically by measuring sugar metabolism (FDG uptake), endothelial permeability (contrast enhancement), and vessel wall thickening. The investigators will also determine whether these changes differ between A-AION and NAION. Furthermore, the investigators aim to study the occurence of subtle retinal changes, particularly paracentral acute middle maculopathy (PAMM) and intra- or subretinal fluid (IRF/SRF), and whether these occur with different frequencies in A-AION compared to NAION.

The study builds on the following hypotheses:

That patients with A-AION show increased FDG uptake, endothelial leakage, and vessel wall thickening in the orbital vessels supplying the eye and optic nerve, as signs of vascular inflammation, and that these changes are not present in NAION.

That GCA patients without vision loss but with signs of orbital vascular inflammation are at increased risk of later vision loss, compared with GCA patients without orbital vascular inflammation.

That subtle retinal changes are common in ischemic optic neuropathy and can function as specific biomarkers to distinguish between A-AION and NAION, thus improving early diagnosis and treatment.

Endpoints:

Substudy 1 (PET/MRI for A-AION vs NAION):

Primary endpoint: FDG uptake, endothelial leakage, and vessel wall thickening in the direct vascular supply of the eye and optic nerve.

Secondary/exploratory endpoints: Correlation with final clinical diagnosis; assessment of FDG uptake and vessel changes in other cranial arteries; characterization of orbital and optic nerve structural changes in NAION.

Substudy 2 (GCA without vision loss):

Primary endpoint: Incidence of ocular complications after 6 months (and possibly again after 2 years) in patients with orbital vascular inflammation versus those without.

Secondary/exploratory endpoints: Frequency and extent of orbital vessel inflammation; occurrence of subclinical structural/functional eye changes and retinal abnormalities (e.g., PAMM, IRF/SRF) in correspondance with orbital vascular inflammation.

Substudy 3 (Retinal biomarkers for A-AION vs NAION):

Primary endpoint: Occurrence of PAMM and IRF/SRF in ischemic optic neuropathy and correlation with the final diagnosis of A-AION versus NAION.

Secondary/exploratory endpoints: Association between retinal abnormalities and orbital inflammation.

Significance:

This study will, to our knowledge, be the first to investigate FDG uptake and endothelial dysfunction in the orbital vessels supplying the eye and optic nerve as markers of inflammation in ischemic optic neuropathy and GCA. It will also be the first large-scale study to examine the relationship between retinal changes (PAMM, IRF/SRF) and final diagnosis of A-AION or NAION.

Results may provide crucial insights into the pathophysiology of ischemic optic neuropathy and GCA, improving diagnostic accuracy and clinical management of both conditions. The findings could help prevent serious complications such as blindness, stroke, or aortic dissection in GCA patients and reduce unnecessary tests and immunosuppressive treatment in NAION patients. Furthermore, by identifying subclinical orbital inflammation, this project may contribute to improved risk stratification and personalized treatment strategies for GCA patients.

Background and literature review:

GCA is a systemic vasculitis affecting large and medium-sized arteries, often associated with polymyalgia rheumatica (PMR), and seen almost exclusively in people over 50. Incidence is highest in Scandinavia, at ~22 cases per 100,000 per year in this age group. Pathogenesis involves an autoimmune response with dysregulated T-cell activation, local dendritic cells, and pro-inflammatory cytokines (IL-1, IL-6, TNF), leading to formation of giant cells, vessel wall damage, and fibrotic remodeling.

Clinically, GCA can cause diverse symptoms, but untreated cases may result in sudden vision loss (A-AION) or systemic complications. Diagnosis is currently based on temporal artery biopsy and imaging methods such as ultrasound (halo and compression signs), MRI (contrast enhancement of vessel walls), and FDG PET (increased uptake in inflamed arteries). Orbital MRI BB has shown subclinical changes, including optic nerve sheath enhancement, in GCA patients without visual symptoms.

OCT imaging has identified ischemic retinal changes such as PAMM and IRF/SRF, which appear to differ between A-AION and NAION. Early data suggest these may serve as highly specific biomarkers for differentiating between the two, but findings require validation in larger, homogeneous cohorts. Since OCT is widely available and non-invasive, validated retinal biomarkers could become essential for rapid diagnosis of ischemic optic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

For AION group:

* Clinical suspicion of newly onset ischemic optic neuropathy (A-AION or NA-AION), defined by ipsilateral findings of: Papilledema; Relevant visual impairment measured by visual acuity and/or visual field; Relative afferent pupillary defect (RAPD), except if mydriatic agents have been administered or if bilateral optic neuropathy is present.
* Age ≥ 50 years

For GCA group:

* Clinically- and ultrasound-confirmed, newly diagnosed GCA
* Absence of visual changes related to GCA in one or both eyes, including: Transient vision loss; permanent vision loss; transient double vision; permanent double vision
* Age ≥ 50 years

Exclusion Criteria:

* Ferromagnetic implants
* Severe renal impairment with eGFR < 30 mL/min/1.73m²
* Allergy to MRI contrast agents
* Severe claustrophobia
* Pregnancy or breastfeeding
* Previously documented ipsilateral optic neuropathy or giant cell arteritis
* More than 5 days of treatment with prednisolone prior to inclusion

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at the Ophthalmological and/or Rheumatological Department at Rigshospitalet, Copenhagen, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2025-11-17 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Orbital vascular inflammation on PET/MRI | 2 years
  To investigate whether there is increased FDG uptake, increased endothelial permeability, and thickening of the vessel wall in the direct vascular supply to the eye and optic nerve, as signs of orbital vascular inflammation, among patients with ischemic optic neuropathy.
Risk of vision loss in GCA | 2 years
  To investigate whether GCA patients without visual symptoms, but with signs of orbital vascular inflammation, have a higher incidence of GCA-related eye disease after 6 months compared to GCA patients without signs of orbital vascular inflammation (and possibly again after 2 years).
Retinal biomarkers in AION | 2 years
  To characterize the occurrence of subtle retinal changes, with a focus on paracentral acute middle maculopathy (PAMM; band-like hyperreflective changes in the middle retinal layers) and intra- and subretinal fluid (IRF/SRF; fluid in or beneath the retina) among patients with ischemic optic neuropathy.

SECONDARY OUTCOMES:
Correlation with final clinical diagnosis | 2 years
  To correlate signs of orbital vascular inflammation with the final clinical diagnosis of GCA / A-AION or NAION.
Occurence of orbital vascular inflammation in GCA without vision loss | 2 years
  To assess the frequency and extent of orbital vascular inflammation among GCA patients without visual symptoms.
Eye examination biomarkers of orbital vascular inflammation | 2 years
  To investigate whether structural or functional eye changes can be detected by neuro-ophthalmological examination (including visual acuity, perimetry, fundus photography, and OCT) in GCA patients without visual symptoms but with orbital vascular inflammation.
Vascular inflammation outside of the orbit | 2 years
  To characterize the occurrence of increased FDG uptake, increased endothelial permeability, and vessel wall thickening, as signs of vascular inflammation, in the walls of other cranial blood vessels among patients with GCA.
Orbital pathophysiologic changes in NAION | 2 years
  To characterize structural and functional changes in the orbit, with a focus on blood vessels and the optic nerve, in patients with NAION.
Retinal biomarkers to diagnose A-AION vs NAION | 2 years
  To correlate the type and frequency of subtle retinal changes with the final clinical diagnosis of A-AION and NAION.

OTHER OUTCOMES:
Pathophysiology behind different retinal biomarkers in AION | 2 years
  To investigate the relationship between the type and degree of retinal changes and the presence of inflammatory and vascular changes in the orbit in patients with A-AION and NAION.